CLINICAL TRIAL: NCT05421403
Title: The Interplay Between Obstructive Sleep Apnea and Inflammatory Cytokines Induces Cognitive Dysfunction in Pediatric Patients
Brief Title: The Interplay Between Obstructive Sleep Apnea Cognitive Dysfunction in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ashraf Wahbaa, Assistant professor of ENT, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUAREC20190509-12
Record Dates: First submitted 2022-06-01; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical (Active Comparator)
  Interventions: Procedure: adenotonsillectomy
- non-Surgical (Placebo Comparator)
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Procedure: adenotonsillectomy — all patients with adenoid or tonsillar or adenotonsillar hypertrophy of grade >2 will undergo adenoidectomy, tonsillectomy or adenotonsillectomy (AT) according to the indication. Overweight or obese patients with mild or moderate OSAS will undergo 6-m trial of lifestyle intervention (LSI) and CPAP if indicated, responders will undergo more follow-up otherwise surgical interference was indicated
  Arms: Surgical
Behavioral: Lifestyle intervention — After baseline testing, all subjects began a structured 6-month LSI consisting of dietary modification and exercise. Intensive dietary counseling was provided weekly for the first 4 weeks of the intervention, monthly subsequently until 6 months. A target caloric deficit of ~250.500 cal/d was recommended throughout dietary counseling. Dietary regimen consisted of diets composed of nutrients contributing to total energy as 55% carbohydrate, 15% protein, and 30% fat. Other lifestyle changes included calorie restriction depending on reduction of the frequency of snack consumption, ingestion of low-calorie and low-fat snacks, limiting sugar-based carbonated drinks and the duration of television watching or mobile games. Exercise sessions consisted of both aerobic and strength training three times weekly.
  Arms: non-Surgical

SUMMARY:
Objectives: Determination of the impact of obstructive sleep apnea (OSA) on the cognitive function (CF) and serum tumor necrosis factor-α (TNF-α), interleukin (IL)-6 and 1β levels in children aged 5-12 years and the effect of OSA management on these variables.

Patients & Methods: 224 patients were evaluated using the Pediatric Sleep Questionnaire, the NEPSY score for CF and Polysomnography (PSG) to grade OSA severity according to the Apnea/hypopnea index (AHI). Patients with adenotonsillar hypertrophy grade >2 will undergo the appropriate surgical intervention. Overweight or obese patients with mild or moderate OSAS will undergo 6-m trial of lifestyle intervention (LSI). Blood samples were obtained for ELISA estimation of cytokines' levels. At end of 6-m follow-up, all variables were re-evaluated

DETAILED DESCRIPTION:
All children aged 5-12 years who attended the outpatient clinics of Otorhinolaryngology and/or Pediatrics with complaints suggestive of OSAS were eligible for evaluation for exclusion and inclusion criteria according to the conditions of the Local Ethical Committee which approved the study protocol by number.

Evaluation Tools

1. Evaluation of body mass index (BMI): BMI was calculated according to Bray as weight (kg) divided by the square height (m2) and was interpreted according to the International Obesity Task Force (IOTF) BMI cut-offs according to the percentile of BMI adjusted for age and gender.
2. Pediatric Sleep Questionnaire (PSQ) using the sleep-related breathing disorders scale which consists of 3 domains including 22 items with three responses to each item Yes (=1), No (=0), and don't know = missed answer.
3. Neurocognitive Assessments using the NEPSY II score which is designed to assess six domains (Appendix 2), each domain was expressed as scaled scores with lower scores indicating cognitive dysfunction.
4. Otorhinolaryngologic assessment variables:

   * Assessment of the volume of the palatine tonsils using Brodsky grading scale Adenoid size was assessed by X-Ray soft tissue nasopharynx lateral view and graded according to. Assessment of the tongue position within the oral cavity to evaluate the extent of obstruction of the oral cavity by the tongue using the modified Mallampati method.
   * Polysomnography (PSG) was performed according to guidelines of the American Academy of Sleep Medicine (AASM) for the scoring of sleep and associated events. The hypopnea index (HI) indicated the number of hypopneas per hour of sleep and the Apnea/hypopnea index (AHI) is the summation of apnea and hypopnea indices.
5. Laboratory investigation: Venous blood samples (5 ml) were collected for ELISA estimation of serum levels of tumor necrosis factor-α (TNF-α), interleukin (IL)-6, and 1β.

Diagnosis and grading of OSAS

1. Diagnosis of OSAS:

   Pediatric OSAS was diagnosed according to guidelines of the American Academy of Sleep Medicine (21) depending on both the clinical findings and the polysomnographic criteria for diagnosis.
2. OSAS severity grading OSAS severity was graded according to the apnea-hypopnea index (AHI) into mild if AHI was 1-4.9, moderate if AHI 5-9.9, or severe if AHI > 10 and if AHI was >30 OSAS is very severe.

ELIGIBILITY:
Inclusion Criteria:

* Children in age range of 5-12 years with mild-to-severe OSAS, free of exclusion criteria were enrolled in the study.

Exclusion Criteria:

* The presence of craniofacial anomalies
* neurological disorders
* very severe OSAS
* OSAS complicated by complex comorbidities
* residual OSAS following adenotonsillectomy (AT), hypothyroidism, or refusal of the suggested therapeutic plans.
* children who failed or were unable to undergo the cognitive function evaluation and those whose parents refused to undergo polysomnography were also excluded from the study.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Relive of OSAS | 6 months
  The effect of relieve of obstruction on sleep-related breathing disorders and cognitive function as judged by the Pediatric Sleep Questionnaire at end of follow up
Effect of weight reduction on sleep-related breathing disorders | 6 months
  The effect of relieve of obstruction and weight reduction on sleep-related breathing disorders as judged by the NESPY score at end of follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Asyut, Egypt